CLINICAL TRIAL: NCT05045469
Title: Therapeutic Effects of Topical Herbal Medicine on Rosacea
Brief Title: Therapeutic Effects of Topical Herbal Medicine -Rhubarb Ointment on Rosacea
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 202101000A3
Record Dates: First submitted 2021-09-07; First posted 2021-09-16 (Actual); Results first posted 2025-04-01 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2024-01

CONDITIONS: Rosacea; Chinese Herbal Medicine
MeSH Terms: conditions — Rosacea

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (dian dao san group) (Active Comparator): Herbal medicine (dian dao san) will be applied to the lesions of rosacea twice a day. Subject will receive persistent treatment for 6 weeks.
  Interventions: Drug: dian dao san
- group B( topical medicine without therapeutic effects) (Placebo Comparator): Placebo (topical medicine without therapeutic effects) will be applied to the lesions of rosacea twice a day. Subject will receive persistent treatment for 6 weeks.
  Interventions: Drug: dian dao san

INTERVENTIONS:
Drug: dian dao san — dian dao san and placebo will be used in the rosacea lesions twice a day for 6 weeks

SUMMARY:
The aim of this study is to investigate the effects of topical herbal medicine in the patients with rosacea.

DETAILED DESCRIPTION:
Rosacea is a chronic inflammatory disorder which affects the cheek, nose, chin, forehead and eyes. It is typically characterized by cutaneous signs such as flushing, erythema, telangiectasia, papules, and pustules in the face. The pathogenic mechanism of rosacea is unknown, and there is no cure for rosacea. The therapeutic approaches include oral medicine, topical medicine and surgical interventions depending on the different subtypes of rosacea. The recent study demonstrates that combination therapy may be more effectively improved the symptoms of rosacea. Dian dao san is a topical herbal compound for reducing the features as flushing, erythema, papules, and pustules for years. The investigators hypothesize that dian dao san can be more beneficial in treating the patients with rosacea and improving the quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Willing to sign inform consent
* Aged above 20 years old with rosacea
* No treatment for rosacea within 2 weeks

Exclusion Criteria:

* With malignant lesion in the rosacea lesion
* Rosacea lesion with high risk of infection
* Allergy to Chinese herbal medicine patch or ointment
* Pregnancy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-08-04 (Actual); Primary Completion 2024-05-23 (Actual); Study Completion 2024-08-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: YUAN-CHIEH YEH, Doctor, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Keelung Chang Gung Memorial Hospital, Keelung, Taiwan

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group A (Dian Dao San Group) | Group B( Topical Medicine Without Therapeutic Effects)
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A (Dian Dao San Group) | Group B( Topical Medicine Without Therapeutic Effects) | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 11 | 23
  >=65 years | 0 | 1 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.08 (14.94) | 52.08 (10.93) | 46.58 (12.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 8 | 18
  Male | 2 | 4 | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants] | 12 | 12 | 24
Region of Enrollment [Number; unit: participants]
  Taiwan | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Reduction of Flushing, Erythema, Telangiectasia, Papules, and Pustules
Description: quantified by Investigator Global Assessment, IGA. IGA is used in the study for assessing the severity of rosacea ranging from 0 (clean) to 4 (most severe).
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group A (Dian Dao San Group) | Group B( Topical Medicine Without Therapeutic Effects)
Number analyzed (Participants) | 12 | 12
score on a scale | 1 (0.43) | 1.92 (0.67)

2. Secondary Outcome: Dermatology Quality of Life Index, DQoL
Description: DQoL is a questionnaire-based scale designed to measure the impact of dermatological conditions on a patient's quality of life. It assesses various aspects, including symptoms, psychological well-being, social activities, and treatment-related effects.
  Scale Range:The DQoL consists of 10 questions, each scored on a scale from 0 to 3:
  0 = Not at all, 1 = A little,2 = A lot,3 = Very much The total score ranges from 0 to 30, where higher scores indicate a greater negative impact of the skin condition on quality of life.
  Interpretation of Scale Scores:
  Total Score 0-1: No or minimal impact; 2-5: Mild impact; 6-10: Moderate impact; 11-20: Significant impact; 21-30: Severe impact Higher DQoL scores indicate worse quality of life due to the skin condition, while lower scores suggest minimal impact.
  Computation of Scores:DQoL total score is calculated as the sum of the 10 item scores.
  Unit of Measure:
  "Scores on a scale" should be used as the Unit of Measure if no other units apply.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group A (Dian Dao San Group) | Group B( Topical Medicine Without Therapeutic Effects)
Number analyzed (Participants) | 12 | 12
score on a scale | 2.83 (2.25) | 6.25 (4.49)

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Group A (Dian Dao San Group) | Group B( Topical Medicine Without Therapeutic Effects)
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-03-12): https://cdn.clinicaltrials.gov/large-docs/69/NCT05045469/Prot_SAP_000.pdf